CLINICAL TRIAL: NCT02662504
Title: Pilot Study of the Feasibility of Intrapleural Photodynamic Therapy in a Multimodal Treatment Combining Extended Pleurectomy/Decortication, Adjuvant Chemotherapy and Prophylactic Radiotherapy in Patients With Malignant Pleural Mesothelioma
Brief Title: Intrapleural Photodynamic Therapy in a Multimodal Treatment for Patients With Malignant Pleural Mesothelioma
Acronym: MesoPDT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); University of Pennsylvania (Other); Région Nord-Pas de Calais, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014_01; 2015-001554-15 (EudraCT Number)
Record Dates: First submitted 2016-01-14; First posted 2016-01-25 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Malignant Pleural Mesothelioma
Keywords: mesothelioma; multimodal treatment; PDT; pleura
MeSH Terms: conditions — Mesothelioma, Malignant; Mesothelioma | interventions — Photochemotherapy; Chemotherapy, Adjuvant; Pemetrexed; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- multimodal treatment + intrapleural PDT (Experimental): * surgery of the MPM: extended pleurectomy/decortication (eP/D)
  * intra-operative (intrapleural) photodynamic therapy (PDT). Briefly, each patient will receive porfimer sodium (PHOTOFRIN®) (2 mg/kg) 24 hours before eP/D (IV injection on 3-5 minutes). Cutaneous light precautions will be instituted immediately and for the next 4 weeks.
  then:
  * prophylactic chest radiotherapy of surgical scars to prevent tumor seeding (3 x 7 Gray)
  * adjuvant standard chemotherapy by (cis)platin 75 mg/m2 and pemetrexed 500 mg/m2 up to 6 cycles (1 cycle every 3 weeks), with oral folic acid (400 μg daily) and vitamin B12 (1000 μg Q9W) supplementation
  Interventions: Device: photodynamic therapy (PDT); Procedure: thoracic surgery Pleurectomy / extended Decortication; Drug: Adjuvant chemotherapy

INTERVENTIONS:
Device: photodynamic therapy (PDT) — Intra-operative (intrapleural) photodynamic therapy (PDT): briefly, each patient will receive porfimer sodium (PHOTOFRIN®) (2 mg/kg) 24 hours before eP/D (IV injection on 3-5 minutes). Cutaneous light precautions will be instituted immediately and for the next 4 weeks.
  After complete macroscopic resection of the tumour, the thoracic surgeon and his team will set isoprobes (7 at least) in the "pleural" cavity to monitor by a dosimetry device the correct illumination of the cavity with a visible red light (wavelength of 630 nm; laser source). PDT-related postoperative considerations include light precautions, intensive focus on perioperative nutrition, and a greater than normal fluid requirement in the immediate postoperative period.
  Other Names: Photofrin
Procedure: thoracic surgery Pleurectomy / extended Decortication — extended P/D is intended to remove any macroscopic tumor including the parietal and visceral pleura when the diaphragm and / or the pericardium was resected
Drug: Adjuvant chemotherapy — Chemotherapy should begin up to three months after surgery. It consists of pemetrexed 500 mg / m2 followed 30 minutes later by cisplatin 75 mg / m2 (in the usual manner from the center to the chemotherapy) on day 1 (J1) of each cycle every 3 weeks, for up to 6 cycles.
  Other Names: pemetrexed / cisplatin

SUMMARY:
Malignant pleural mesothelioma (MPM) is an aggressive tumour with poor prognosis (median survival <13 months), and high resistance to chemotherapy. Extended pleurectomy/decortication (eP/D) is a debulking surgery of MPM but cannot be considered as a curative treatment. Therefore it has been suggested that eP/D may be of interest if combined with intra-operative treatment and adjuvant therapies.

Photodynamic Therapy (PDT) is an innovative treatment based on the rationale that tumour cells, if previously treated with photosensitizing drugs (Photofrin), will die when exposed to light at a particular wavelength. Interestingly PDT might also stimulate anti-tumour immune response through the release of tumour antigens and induced inflammation.

PDT was tested in phase I-II trials for MPM in combination with EPP or eP/D, and chemotherapy. US studies from J Friedberg et al found very promising survival results in MPM when combining eP/D, but not EPP, intra-operative PDT and chemotherapy (cisplatin-pemetrexed), with a median overall survival of 31.7 months.

However, the definitive value of intra-pleural PDT combined to eP/D in the treatment of MPM still need to be validated. The same multimodal treatment has been established in Lille, the French national expert centre for MPM, with the help of our american colleagues. Therefore, this phase II trial proposes to patients to benefit from the combination of eP/D, intra-operative PDT then chemotherapy by cisplatin-pemetrexed and prophylactic radiotherapy.

Primary endpoint is the feasibility for the patients to have the full multimodal treatment of MPM including intrapleural PDT without unacceptable or unexpected grade III-IV toxicities. Secondary endpoints are PFS, OS, ORR, and quality of life. If the feasibility of such treatment would be confirmed in France, a multicentric, randomized trial comparing this experimental treatment vs control arm (same multimodal treatment without PDT) is planned.

DETAILED DESCRIPTION:
phase II trial assessing the feasibility of an experimental multimodal treatment combining:

* surgery of the MPM: extended pleurectomy/decortication (eP/D)
* intra-operative (intrapleural) photodynamic therapy (PDT). Briefly, each patient will receive porfimer sodium (PHOTOFRIN®) (2 mg/kg) 24 hours before eP/D (IV injection on 3-5 minutes). Cutaneous light precautions will be instituted immediately and for the next 4 weeks.

then:

* prophylactic chest radiotherapy of surgical scars to prevent tumor seeding (3 x 7 Gray)
* adjuvant standard chemotherapy by (cis)platin 75 mg/m2 and pemetrexed 500 mg/m2 up to 6 cycles (1 cycle every 3 weeks), with oral folic acid (400 μg daily) and vitamin B12 (1000 μg Q9W) supplementation
* follow-up

ELIGIBILITY:
Inclusion Criteria:

* histologically-proved epithelioid malignant pleural mesothelioma (MPM) on biopsies obtained before eP/D surgery
* tumor stage: no tumor extension to controlateral lung, mediastinum, peritoneum or myocardium (<T4); mediastinal lymph nodes extension: cN2 but no bulky N2 or N3), no metastasis (M0)
* Performance status WHO PS 0-1
* patients fit to have surgery (eP/D) and chemotherapy (cisplatin-pemetrexed), based on clinical examination, complete normal biological work-up, full assessment by cardiac and pulmonary function tests. Predicted post-surgical values should be sufficient for normal daily life: FEV1>40%; pre-surgical DLCO>50% predicted value and VO2max >15 ml/min/kg; (left ventricular) cardiac function >50% and no significant pulmonary artery hypertension
* written informed consent must be obtained before inclusion and randomization

Exclusion Criteria:

* Another histologic subtype than epithelioid MPM at the time of diagnosis
* Bulky N2, N3 and/or M1 stage (UICC/IMIG 1995)
* prior chemotherapy for mesothelioma
* prior radiotherapy of thorax, neck or upper abdomen
* other malignancy treated within 5 years, except basal cell carcinoma or in situ carcinoma of the cervix
* contra-indication for MPM surgery or chemotherapy (cisplatin and pemetrexed): cardiac failure, pulmonary hypertension, liver or kidney dysfunction (GFR<60 ml/min), uncontrolled infection, previous major neurotoxicity or ototoxicity,... or other severe condition according to the investigator
* pregnancy or breast feeding
* contra-indication for porfimer sodium (Photofrin): porphyria or known hypersensitivity to porphyrins, severe hepatic impairment, tracheo-oesophageal or broncho-oesophageal fistula, suspected erosion of major blood vessels due to risk of massive, potentially fatal haemorrhage
* A previous talc pleurodesis during diagnostic thoracoscopy is NOT an exclusion criteria but talc on mediastinal pleura should be avoided to not keep away from eP/D.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-01-16 (Actual); Primary Completion 2018-03-12 (Actual); Study Completion 2018-03-13 (Actual)

PRIMARY OUTCOMES:
Number of Patients having the full multimodal treatment without unacceptable and unexpected toxicities (grade ≥ 3) graded According to NCI CTC Version 4.0 | at 12 months

SECONDARY OUTCOMES:
Number of responders or stable patients after surgery | at 12 months
Progression-free survival (PFS) | through study completion, an average of 13 months
Quality of life assessed by a specific questionnaire MPM (HCCA EORTC-30) | Baseline and at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Scherpereel, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- CHRU de Lille Hôpital Calmette, Lille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Munck C, Mordon S, Betrouni N. Illumination profile characterization of a light device for the dosimetry of intra-pleural photodynamic therapy for mesothelioma. Photodiagnosis Photodyn Ther. 2016 Dec;16:23-26. doi: 10.1016/j.pdpdt.2016.08.010. Epub 2016 Sep 1. PMID 27594672